CLINICAL TRIAL: NCT03705286
Title: Randomized Trial of Endotracheal Tubes to Prevent Ventilator-Associated Pneumonia - PreVent 2 Study
Brief Title: Endotracheal Tubes to Prevent Ventilator-Associated Pneumonia
Acronym: PreVent2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Miriam Treggiari, Professor, Vice Chair of Clinical Research, Anesthesiology, Yale University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2000027877; R33HL138650 (NIH)
Record Dates: First submitted 2018-10-03; First posted 2018-10-15 (Actual); Results first posted 2024-09-24 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Ventilator-acquired Pneumonia
Keywords: Pneumonia; Endotracheal intubation
MeSH Terms: conditions — Pneumonia, Ventilator-Associated; Pneumonia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- PVC-ETT (Active Comparator): Polyvinylchloride endotracheal tube
  Interventions: Device: PVC-ETT
- EVAC-PU-ETT (Experimental): Continuous aspiration of subglottic secretions with polyurethane cuff endotracheal tube
  Interventions: Device: EVAC-PU-ETT

INTERVENTIONS:
Device: EVAC-PU-ETT — Placement of a EVAC-PU-ETT in the setting of emergent intubation.
  Other Names: Shiley™ Evac Oral Tracheal Tube, SealGuard™, Murphy Eye
  Arms: EVAC-PU-ETT
Device: PVC-ETT — Placement of a PVC-ETT in the setting of emergent intubation.
  Other Names: Shiley™ Cuffed Basic Endotracheal Tube
  Arms: PVC-ETT

SUMMARY:
Researchers are looking at two different types of breathing tubes to see if one is better than the other at preventing pneumonia. One of the tubes has a design features to prevent leakage of fluids from the mouth and the back of the throat into the lower airways and lungs. This is important since leakage of small amounts of fluid into the lungs may lead to pneumonia. The other tube is the standard tube used at most hospitals.

The hypothesis is that the use of a breathing tube that reduces fluid leakage into the lungs will reduce the risk of developing pneumonia and improve quality of life and cognitive function, compared to the standard tube. The study will also look at the safety of the modified breathing tube, compared to the standard tube.

DETAILED DESCRIPTION:
The proposed study will be a randomized, controlled trial, conducted under Exception From Informed Consent (EFIC), comparing patients who undergo emergency tracheal intubation with one of two different endotracheal tubes (ETTs), one of which is designed to prevent ventilator-associated pneumonia (VAP): 1) An ETT fitted with a lumen to allow continuous aspiration of subglottic secretions and made with a polyurethane cuff (EVAC-PU-ETT); and 2) A standard ETT with a polyvinylchloride cuff (PVC-ETT). Approximately 1,074 adult patients requiring endotracheal intubation in the ED or hospital for acute respiratory distress or failure will be randomly assigned in an equal fashion to be intubated with one of the two ETTs (537 patients in each group). Because endotracheal intubation is performed in an emergency setting, the unit of randomization will be the intubation kits containing, in a concealed manner, one of the two types of ETT. The intubation kits are placed in areas where emergency intubation teams receive their intubation equipment supplies, primarily in the ICUs and in the emergency department. The study is designed to allow all patients requiring emergency intubation to be potentially eligible for enrollment to ensure the applicability of the study findings to a generalizable setting of patients receiving emergency intubation outside the operating room.

The trial primary aim is to determine if EVAC-PU-ETT is as safe as PVC-ETT and if long-term patient quality of life and cognitive function are better in PU-CASS-ETT, compared with PVC-ETT. The investigators will also monitor any device-related adverse events. Additional secondary endpoints include the incidence of infection-related ventilator associated conditions (IVAC) and ventilator associated events (VAEs), as defined by the Center for Disease Control, respiratory antibiotics use, incidence of "clinical" VAP, 28-day ventilator-free days, mean daily Sequential Organ Failure Assessment (SOFA) score, length of ICU and hospital stay, and mortality up to six months will serve to evaluate other clinical meaningful consequences resulting from the occurrence of VAP. Furthermore, the study will perform economic evaluation (cost-consequence approach) of quality of life, healthcare resource utilization and cost for hospitals. Primary and secondary endpoints will be compared between the PU-CASS-ETT and PVC-ETT groups, using an intention-to-treat approach.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years of age
2. Requiring emergency endotracheal intubation in the ED or in-hospital for acute respiratory distress or failure
3. A study intubation kit containing the study ID number must have been used for the emergency intubation
4. Admitted to the ICU and receiving mechanical ventilation

Exclusion Criteria:

1. Patients electively intubated in the operating room whether or not they require subsequent ICU admission
2. Use of a non-study designated intubation kit (such as nasal intubation, tracheotomy, intubation occurring at a location not supplied with the study intubation kits)
3. Patients with permanent tracheostomy
4. Protected populations including children (age <18 years), pregnant women, or prisoners
5. Evidence of unwillingness to participate in a research study as documented in the patient's electronic health record, or at the time of intubation if there is opportunity to read the opt-out script.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1074 (Actual)
Dates: Start 2019-05-06 (Actual); Primary Completion 2023-02-23 (Actual); Study Completion 2023-02-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Miriam M Treggiari, MD, PhD, MPH, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Treggiari MM, Sharp ES, Ohnuma T, Fajardo EC, Aydin A, Akhtar S, Kampp M, Hashemaghaie M, Potnis A, Gugel T, Simon J, Curry LG, Adams K, Darji B, Sureshanand S, Hintz R, Lorzano SN, Johnson C, Yanez ND. Hospital and long-term outcomes for subglottic suction and polyurethane cuff versus standard endotracheal tubes in emergency intubation (PreVent 2): a randomised controlled phase 2 trial. Lancet Respir Med. 2025 Nov 27:S2213-2600(25)00294-2. doi: 10.1016/S2213-2600(25)00294-2. Online ahead of print. PMID 41319662

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 4 patients inadvertently enrolled; 2 patients refused continued participation
Period: Overall Study
Arm/Group | PVC-ETT | EVAC-PU-ETT
Started | 533 | 535
Completed | 87 | 70
Not Completed | 446 | 465

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PVC-ETT | EVAC-PU-ETT | Total
Number analyzed (Participants) | 533 | 535 | 1068
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.6 (15.4) | 63.1 (16.1) | 62.9 (15.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 201 | 196 | 397
  Male | 332 | 339 | 671
Race (NIH/OMB) [Count of Participants; unit: Participants] — 'More than one' racial category was not collected.
  Participants
    American Indian or Alaska Native | 1 | 2 | 3
    Asian | 14 | 8 | 22
    Native Hawaiian or Other Pacific Islander | 2 | 3 | 5
    Black or African American | 102 | 100 | 202
    White | 359 | 359 | 718
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 55 | 63 | 118

OUTCOME MEASURES:

1. Primary Outcome: Quality of Life - 36-item Short-Form General Health Survey
Description: Physical Component Score and Mental Component Score each have scores that range from 0 - 100; Lower scores = more disability, higher scores = less disability.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PVC-ETT | EVAC-PU-ETT
Number analyzed (Participants) | 69 | 84
score on a scale
  Physical Component Score | 40.5 (11.9) | 40.0 (13.1)
  Mental Component Score | 48.9 (12.2) | 45.9 (13.1)
Statistical Analysis 1: Comparison: PVC-ETT vs EVAC-PU-ETT; We evaluated whether there are differences in the Physical Component Score (PCS) for QOL between the PU-EVAC and PVC treatment groups by comparing their respective mean scores (i.e., mean[PU-EVAC] - mean[PVC] ). We modeled the data using linear regression and used robust standard error estimates to construct our statistical test and 95% confidence interval estimates. We also estimated the treatment groups' mean quality of life scores with standard error estimates and 95% confidence intervals; Test type: Superiority; p = 0.78, Regression, Linear; Mean Difference (Final Values) = -0.52, 95% CI 2-sided [-4.21 to 3.17], Standard Error of Mean 1.87
Statistical Analysis 2: Comparison: PVC-ETT vs EVAC-PU-ETT; We evaluated whether there are differences in the Mental Component Score (MCS) for QOL between the PU-EVAC and PVC treatment groups by comparing their respective mean scores (i.e., mean[PU-EVAC] - mean[PVC] ). We modeled the data using linear regression and used robust standard error estimates to construct our statistical test and 95% confidence interval estimates. We also estimated the treatment groups' mean quality of life scores with standard error estimates and 95% confidence intervals; Test type: Superiority; p = 0.15, Regression, Linear; Mean Difference (Final Values) = -2.98, 95% CI 2-sided [-7.03 to 1.07], Standard Error of Mean 2.05

2. Primary Outcome: Cognitive Function
Description: Percentage of patients cognitively impaired, assessed by the National Alzheimer Coordinating Center's Uniform Data Set
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | PVC-ETT | EVAC-PU-ETT
Number analyzed (Participants) | 67 | 82
Participants | 54 | 70
Statistical Analysis 1: Comparison: PVC-ETT vs EVAC-PU-ETT; Test type: Superiority; p = 0.05, Regression, Logistic; Risk Difference (RD) = 0.05, 98% CI 2-sided [-0.07 to 0.17]

3. Secondary Outcome: Airway Related Complications
Description: The number of participants that experienced airway related adverse events.
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | PVC-ETT | EVAC-PU-ETT
Number analyzed (Participants) | 70 | 86
participants | 49 | 71
Statistical Analysis 1: Comparison: PVC-ETT vs EVAC-PU-ETT; We evaluated whether there are differences in the risk of laryngeal injury between the PU-EVAC and PVC treatment groups, comparing their respective risk difference (i.e., probability[PU-EVAC] - probability [PVC]). We fit a logistic regression model and incorporated robust (i.e., Huber-White heteroskedastic consistent) standard error estimates for our hypothesis test and 95% confidence interval estimates; Test type: Superiority; p = 0.05, Regression, Logistic; Risk Difference (RD) = 0.126, 95% CI 2-sided [-0.01 to 0.26]

ADVERSE EVENTS:
Time Frame: up to 6 months
Description: These are all adverse events that were collected during the hospitalization period.
Arm/Group | PVC-ETT | EVAC-PU-ETT
All-Cause Mortality (participants affected / at risk) | 284/533 | 274/535
Serious Adverse Events (participants affected / at risk) | 0/533 | 0/535
Other Adverse Events (participants affected / at risk) | 49/533 | 71/535
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | PVC-ETT (N=533) | EVAC-PU-ETT (N=535)
Cuff leak (Product Issues) | 2 (2) | 6 (6)
Orophrayngeal injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Unplanned extubation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cuff under-inflated (Product Issues) | 1 (1) | 1 (1)
Cuff rupture (Product Issues) | 2 (2) | 0 (0)
Pilot balloon damage (Product Issues) | 2 (2) | 3 (3)
ETT connection mulfunction (Product Issues) | 1 (1) | 0 (0)
Failed extubation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Airway Related Complications (Respiratory, thoracic and mediastinal disorders) | 49/70 (49) | 71/86 (71)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-06-23): https://cdn.clinicaltrials.gov/large-docs/86/NCT03705286/Prot_SAP_000.pdf
  • Informed Consent Form (2020-08-31): https://cdn.clinicaltrials.gov/large-docs/86/NCT03705286/ICF_001.pdf